CLINICAL TRIAL: NCT02316860
Title: The Diagnostic Performance of Tilt Test in Athletes and a Novel Strategy for Its Improvement
Brief Title: The Diagnostic Performance of Tilt Test in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine-Cardiologist, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sportscardiology
Record Dates: First submitted 2014-12-06; First posted 2014-12-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- History of reflex syncope (Other): Passive tilt test in athletes with a history of reflex syncope
  Interventions: Other: Passive tilt test
- No history of reflex syncope (Other): Passive tilt test in athletes without history of reflex syncope
  Interventions: Other: Passive tilt test

INTERVENTIONS:
Other: Passive tilt test — Passive tilt test (without pharmacological provocation). After a horizontal supine rest period of 5 min, the tilt table was inclined at 60° head-up position for 30 min. A positive response was defined according to the European Society of Cardiology guidelines for the diagnosis and management of syncope

SUMMARY:
In the present study the investigators evaluate the sensitivity and specificity of passive tilt test in athletes, as well as their haemodynamic responses and autonomic nervous system activity during head-up tilt. Moreover, the investigators try to apply a novel algorithm for the improvement of diagnostic yield of tilt test in athletes.

DETAILED DESCRIPTION:
We examine athletes with a history of reflex syncope and athletes without history of reflex syncope.All subjects undergo a tilt test, for the evaluation of haemodynamics, heart rate variability (HRV) and baroreflex sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 14-40 years old,
* more than 5 years of exercise training experience and competition at a regional level at different sports

Exclusion Criteria:

* smoking,
* recent alcohol consumption,
* presence of any chronic disease and use of drugs

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of tilt test in athletes as measured by the occurence of syncope/presyncope during tilt test | 30 min
  sensitivity = number of subjects with syncope/presyncope during tilt test/ number of subjects with a history of reflex syncope, specificity = number of subjects without syncope/presyncope during tilt test/ number of subjects without history of reflex syncope

SECONDARY OUTCOMES:
Parameters of haemodynamics during tilt test | 30 min
  We investigate whether the mean values of parameters of haemodynamics during tilt test can discriminate between athletes with a history of reflex syncope and those without history of syncope
Parameters of heart rate variability during tilt test | 30 min
  We investigate whether the mean values of parameters of heart rate variability during tilt test can discriminate between athletes with a history of reflex syncope and those without history of syncope
Parameters of baroreflex sensitivity during tilt test | 30 min
  We investigate whether the mean values of parameters of baroreflex sensitivity during tilt test can discriminate between athletes with a history of reflex syncope and those without history of syncope

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Kouidi, Professor, Principal Investigator — Laboratory of Sports Medicine, Sports Medicine Division, Aristotle University of Thessaloniki, Thessaloniki, Greece
Locations (1):
- Laboratory of Sports Medicine, Sports Medicine Division, Aristotle University of Thessaloniki, Thessaloniki, Greece, Thessaloniki, Greece